CLINICAL TRIAL: NCT00444951
Title: Evaluation of the Response to a Single Dose of Menactra® in Adolescents Aged 16 to 19 Years Who Previously Received One Dose of Quadrivalent (A, C, Y, W 135) and at Least One Dose of Bivalent (A, C) Meningococcal Polysaccharide Vaccine in Saudi Arabia.
Brief Title: Immunogenicity and Safety of Menactra® Vaccine in Adolescents in Saudi Arabia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MTA40
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Results first posted 2011-03-04 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-06

CONDITIONS: Neisseria Meningitidis; Meningococcal Infections
Keywords: N meningitidis
MeSH Terms: conditions — Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Menactra® group (Experimental): Have received previously a dose of an A, C, Y, W 135 and at least one dose of bivalent A, C meningococcal polysaccharide vaccine, will receive a booster dose of Menactra® (Meningococcal [serogroups A, C, Y, W-135] polysaccharide diphtheria toxoid conjugate) vaccine.
  Interventions: Biological: Menactra®: Meningococcal A, C, Y, and W 135 Polysaccharide Diphtheria Toxoid Conjugate vaccine
- Mencevax® group (Experimental): Have received previously a dose of an A, C, Y, W 135 and at least one dose of bivalent A, C meningococcal polysaccharide vaccine, will receive a booster dose of Mencevax ACWY (serogroups A, C, Y, W-135) polysaccharide meningococcal vaccine.
  Interventions: Biological: Mencevax®: Group A, C, W135 and Y polysaccharide meningococcal vaccine
- Control group (Experimental): Participants have not previously received any meningococcal vaccine, will receive a booster dose of Menactra® (Meningococcal [serogroups A, C, Y, W-135] polysaccharide diphtheria toxoid conjugate) vaccine.
  Interventions: Biological: Menactra®: Meningococcal A, C, Y, and W 135 Polysaccharide Diphtheria Toxoid Conjugate vaccine

INTERVENTIONS:
Biological: Menactra®: Meningococcal A, C, Y, and W 135 Polysaccharide Diphtheria Toxoid Conjugate vaccine — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Menactra® group
Biological: Mencevax®: Group A, C, W135 and Y polysaccharide meningococcal vaccine — 0.5 mL, Subcutaneous
  Other Names: Mencevax®
  Arms: Mencevax® group
Biological: Menactra®: Meningococcal A, C, Y, and W 135 Polysaccharide Diphtheria Toxoid Conjugate vaccine — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Control group

SUMMARY:
This study will be conducted among adolescents in Saudi Arabia who previously received one dose of A, C, Y, W 135 and at least one dose of A, C meningococcal polysaccharide vaccine. This study will evaluate the booster administration of Menactra® (Meningococcal A, C, Y, and W 135 Polysaccharide Diphtheria Toxoid Conjugate vaccine) compared with Mencevax® (Meningococcal A, C, Y, and W 135 Polysaccharide vaccine)in terms of their serum bactericidal antibody responses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, as determined by medical history and physical examination.
* Aged between 16 to 19 years on the day of inclusion (from 16th birthday to 1 day before 20th birthday inclusive).
* For the Menactra® and Mencevax® groups, one dose of quadrivalent (A, C, Y, W 135) and at least one dose of bivalent (A, C) meningococcal polysaccharide vaccine with no meningococcal vaccine received less than 2 years prior to enrollment.
* For the Control group, no previous history of any meningococcal vaccination.
* Informed consent form signed by the parent(s) or other legal representative for subject under 18 years and signed by subject him/herself if subject above 18 years old
* Able to provide a vaccination log or has available vaccination record in the Health Center
* Able to attend all scheduled visits and to comply with all trial procedures

Exclusion Criteria:

* Serious chronic disease (i.e., cardiac, renal, neurologic, metabolic, rheumatologic, psychiatric, etc.)
* Known or suspected impairment of immunologic function.
* Acute medical illness with or without fever within the last 72 hours or an oral temperature ≥ 37.5°C at the time of inclusion.
* Administration of immune globulin or other blood products within the last three months, injected or oral corticosteroids or other immunomodulatory therapy within six weeks of the study vaccine. Individuals on a tapering dose schedule of oral steroids lasting < 7 days may be included in the trial provided that they have not received more than one course within the last two weeks prior to enrollment.
* Oral or injected antibiotic therapy within the 72 hours prior to vaccination
* Received any vaccine in the 14-day period prior to study vaccination, or scheduled to receive any vaccination during the 14-day period after study vaccination.
* Previous history of documented invasive meningococcal disease.
* Systemic hypersensitivity to any of the vaccines components or history of a life-threatening reaction to the trial vaccines or a vaccine containing the same substances
* Participation in another clinical trial in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Any condition, which, in the opinion of the investigator, would pose a health risk to the subject, or interfere with the evaluation of the vaccine.
* Personal or family history of Guillain Barré syndrome.
* For female, known or suspected to be pregnant at the time of inclusion

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 450 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc
Locations (7):
- Saudi Arabia (7):
  - AlKhaleej, Al-Qassim Region
  - AlRabwa, Al-Qassim Region
  - S. Buraida, Al-Qassim Region
  - Safra-Al Midhnab, Al-Qassim Region
  - Helal Ahmar, Mecca Region
  - Iskan, Mecca Region
  - Mecca, Mecca Region

REFERENCES:
- [Background] Khalil M, Al-Mazrou Y, Findlow H, Chadha H, Bosch Castells V, Oster P, Borrow R. Meningococcal serogroup C serum and salivary antibody responses to meningococcal quadrivalent conjugate vaccine in Saudi Arabian adolescents previously vaccinated with bivalent and quadrivalent meningococcal polysaccharide vaccine. Vaccine. 2014 Sep 29;32(43):5715-21. doi: 10.1016/j.vaccine.2014.08.026. Epub 2014 Aug 20. PMID 25151042
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 17 February 2007, to 01 July 2007, in 7 clinic centers in Saudi Arabia.
Pre-assignment Details: A total of 450 participants who met the inclusion and exclusion criteria were enrolled, and 446 were vaccinated.
Groups:
- Menactra® Group: Participants have received previously a dose of an A, C, Y, W-135 vaccine and at least one dose of bivalent A, C meningococcal polysaccharide vaccine, received a booster dose of Menactra® (Meningococcal [serogroups A, C, Y, W-135] polysaccharide diphtheria toxoid conjugate) vaccine.
- Mencevax® Group: Participants who had previously been given 1 dose of quadrivalent (A, C, Y, W-135) and at least 1 dose of bivalent (A, C) meningococcal polysaccharide vaccine received a booster dose of Mencevax ACWY (serogroups A, C, Y, W-135) polysaccharide meningococcal vaccine.
- Control Group: Participants who had not previously been given any meningococcal vaccine received 1 dose of Menactra®, meningococcal (serogroups A, C, Y, W-135) polysaccharide diphtheria toxoid conjugate vaccine.
Period: Overall Study
Arm/Group | Menactra® Group | Mencevax® Group | Control Group
Started | 145 | 142 | 163
Completed | 140 | 136 | 160
Not Completed | 5 | 6 | 3
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menactra® Group | Mencevax® Group | Control Group | Total
Number analyzed (Participants) | 145 | 142 | 163 | 450
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 110 | 115 | 134 | 359
  Between 18 and 65 years | 35 | 27 | 29 | 91
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 17.90 (1.20) | 17.77 (1.15) | 17.85 (1.15) | 17.84 (1.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 78 | 53 | 209
  Male | 67 | 64 | 110 | 241
Region of Enrollment [Number; unit: participants]
  Saudi Arabia | 145 | 142 | 163 | 450

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Vaccine Serogroups Determined by Serum Bactericidal Activity Using Baby Rabbit Complement (SBA-BR) Pre- and Post-Menactra® Vaccination
Time Frame: Baseline (Day 0) and Day 28 after vaccination
Population: Geometric mean titers were evaluated in participants who received vaccine injection (full analysis set population).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dil)
Arm/Group | Menactra® Group | Mencevax® Group | Control Group
Number analyzed (Participants) | 144 | 141 | 161
Titers (1/dil)
  Serogroup A (Baseline) | 651.5 [496.4 to 854.9] | 889.7 [699.5 to 1131.5] | 441.1 [327.8 to 593.4]
  Serogroup A (Day 28) | 4116.3 [3468.7 to 4884.9] | 3833.4 [3308.4 to 4441.7] | 6351.6 [5508.3 to 7324.0]
  Serogroup C (Baseline) | 14.7 [9.9 to 22.0] | 15.8 [10.4 to 23.8] | 16.8 [11.1 to 25.4]
  Serogroup C (Day 28) | 288.3 [190.2 to 437.0] | 158.6 [99.7 to 252.0] | 993.4 [714.5 to 1381.2]
  Serogroup Y (Baseline) | 78.8 [49.7 to 125.0] | 73.4 [44.7 to 120.7] | 16.8 [11.1 to 25.3]
  Serogroup Y (Day 28) | 2770.1 [2197.0 to 3492.6] | 1936.3 [1425.7 to 2629.8] | 4204.6 [3458.2 to 5112.0]
  Serogroup W-135 (Baseline) | 18.5 [11.8 to 29.0] | 24.5 [15.2 to 39.6] | 8.1 [5.6 to 11.8]
  Serogroup W-135 (Day 28) | 2435.5 [1714.7 to 3459.3] | 1455.7 [958.1 to 2211.7] | 6926.7 [5647.9 to 8495.1]

2. Secondary Outcome: Percentage of Participants With At Least a 4-Fold Rise in Titers Determined by Serum Bactericidal Activity Using Baby Rabbit Complement (SBA-BR) Post-Menatcra® Vaccination
Time Frame: Baseline (Day 0) and Day 28 After Vaccination
Population: 4-Fold rise titers were determined in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Menactra® Group | Mencevax® Group | Control Group
Number analyzed (Participants) | 140 | 136 | 160
Percentage of Participants
  Serogroup A | 66 | 62 | 86
  Serogroup C | 71 | 57 | 81
  Serogroup Y | 80 | 69 | 96
  Serogroup W-135 | 84 | 72 | 96

3. Secondary Outcome: Number of Participants Reporting a Solicited Injection Site or Systemic Reactions Post-vaccination
Time Frame: Day 0 to Day 7 Post-vaccination
Population: Safety analysis was on all vaccinated participants, intend-to-treat population (Safety analysis set)
Measure: Number; unit: Participants
Arm/Group | Menactra® Group | Mencevax® Group | Control Group
Number analyzed (Participants) | 144 | 141 | 160
Participants
  Any Solicited Injection Site Reaction | 88 | 71 | 98
  Any Injection Site Pain | 85 | 66 | 95
  Grade 3 Injection Site Pain (Incapacitating) | 10 | 3 | 9
  Any Injection Site Erythema | 39 | 34 | 42
  Grade 3 Injection Site Erythema (≥ 5 cm) | 0 | 1 | 2
  Any Injection Site Swelling | 46 | 29 | 34
  Grade 3 Injection Site Swelling (≥ 5 cm) | 0 | 0 | 4
  Any Solicited Systemic Reaction | 87 | 86 | 90
  Any Fever | 25 | 17 | 16
  Grade 3 Fever (> 39.0 ºC) | 3 | 1 | 0
  Any Headache | 66 | 64 | 60
  Grade 3 Headache (Prevents daily activities) | 8 | 6 | 8
  Any Malaise | 61 | 55 | 61
  Grade 3 Malaise (Prevents daily activities) | 8 | 7 | 6
  Any Myalgia | 60 | 55 | 72
  Grade 3 Myalgia (Prevents daily activities) | 10 | 8 | 10

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 to 1 month post-vaccination
Arm/Group | Menactra® Group | Mencevax® Group | Control Group
Serious Adverse Events (participants affected / at risk) | 1/144 | 0/141 | 0/160
Other Adverse Events (participants affected / at risk) | 85/144 | 66/141 | 95/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Menactra® Group (N=144) | Mencevax® Group (N=141) | Control Group (N=160)
Perianal abcess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Menactra® Group (N=144) | Mencevax® Group (N=141) | Control Group (N=160)
Injection site pain (General disorders) | 85/142 (85) | 66/138 (66) | 95/158 (95)
Injection site erythema (General disorders) | 39/142 (39) | 34/138 (34) | 42/158 (42)
Injection site swelling (General disorders) | 46/142 (46) | 29/138 (29) | 34/158 (34)
Fever (General disorders) | 25/142 (25) | 17/138 (17) | 16/158 (16)
Headache (Nervous system disorders) | 66/142 (66) | 64/138 (64) | 60/158 (60)
Malaise (Gastrointestinal disorders) | 61/142 (61) | 55/138 (55) | 61/158 (61)
Myalgia (Musculoskeletal and connective tissue disorders) | 60/142 (60) | 55/138 (55) | 72/158 (72)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.